CLINICAL TRIAL: NCT05493033
Title: A Multicenter Randomized Clinical Trial Comparing Intracorporeal and Extracorporeal Ileocolic Anastomotic After Laparoscopic Right Colectomy for Colon Cancer (COLOR IV)
Brief Title: Intracorporeal Versus Extracorporeal Anastomotic After Laparoscopic Right Colectomy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, Zhongtao Zhang, professor, Beijing Friendship Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COLOR IV Trial
Record Dates: First submitted 2022-05-23; First posted 2022-08-09 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Colon Cancer
Keywords: laparoscopic; intracorporeal anastomosis; anastomotic leak
MeSH Terms: conditions — Colonic Neoplasms; Anastomotic Leak

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intracorporeal anastomotic after LRC (Experimental)
  Interventions: Procedure: Intracorporeal anastomotic after LRC
- Extracorporeal anastomotic after LRC (Active Comparator)
  Interventions: Procedure: Extracorporeal anastomotic after LRC

INTERVENTIONS:
Procedure: Intracorporeal anastomotic after LRC — Complete laparoscopic dissection of the mesocolon is mandatory. D2 or D3/CME is optional. And the extent of colon resection is based on the location of the tumor while the ileocecal resection is excluded. After fully mobilization of the colon and mesentery, the terminal ileum and transverse colon will be transected by a laparoscopic linear stapler. The side-to-side anastomosis is performed laparoscopically. The enterotomy is closed by a double-layer suture. All the anastomotic procedures are completed laparoscopically. The specimen is then removed through a Pfannenstiel incision within a specimen bag.
  Arms: Intracorporeal anastomotic after LRC
Procedure: Extracorporeal anastomotic after LRC — The procedures of the mobilization and vessel ligation are similar. After that, the mobilized colon and terminal ileum are brought out through the upper mid-line incision with the wound protector. The colon and terminal ileum are similarly dissected distally to the specimen with a stapling device. The side-to-side anastomosis is completed and the anastomotic site is reinforced. The anastomotic bowel is returned to the abdominal cavity.
  Arms: Extracorporeal anastomotic after LRC

SUMMARY:
Background: Laparoscopic assisted right hemicolectomy is recommended for right colon cancer. As a more minimally invasive procedure, intracorporeal ileocolic anastomosis has potential advantages: reducing torsion and traction on the mesentery, reducing skin incision length and enhancing postoperative recovery. However, the longer operative time, greater risk of intra-abdominal infection and steep learning curve for intestinal anastomosis performed under laparoscopic conditions, does this increase the incidence of postoperative complications, especially the incidence of anastomotic leakage, and whether it affects There is no high-level research evidence on the survival of patients.

Study design: COlOR IV study is an international prospective, multicenter, randomized controlled clinical study of intraperitoneal anastomosis versus extraperitoneal anastomosis after laparoscopic right hemicolectomy for colon cancer . The study will include a quality assessment phase before randomisation to ensure required competency level and uniformity of the intracorporeal and extracoporeal techniques.

Endpoint: Primary outcome is anastomotic leakage within 30 days after surgery. Main secondary endpoint is 3-year disease-free survival rate. Secondary endpoints are mortality and morbidity, postoperative recovery, overall survival, surgical specimen quality, quality of life.

Statistics: The primary endpoint is anastomotic leakage within 30 days after surgery. The anastomotic leakage rate was set to 2% in the both groups, and an increase in the incidence of anastomotic leakage of 2.5% was considered inferior. The one-sided significance level was 0.025, the power was 0.9. The dropout rate was 20%, and taking into account the post-randomization analysis (dropout 5%), the total sample size was 1158. There were 579 cases in the intracorporeal anastomosis group and 579 cases in the extracorporeal anastomosis group.

Main selection: Patients with histologically proven right colon cancer (cecum, ascending colon and proximal 1/3 of the transverse colon malignant tumor), clinically stage I-III, and intention for right hemicolectomy with primary anastomosis.

Hypothesis: The hypothesis is that intracoporeal anastomosis will have comparable anastomotic leak rate and 3-year DFS, but faster postoperative recovery with extracoporeal anastomosis.

ELIGIBILITY:
Inclusion criteria

1. Age: 18 ~ 80 years, male or female;
2. Histological or cytological diagnosis of right colon cancer (cecum, ascending colon and proximal 1/3 of the transverse colon cancer);
3. Stage I-III according to the AJCC-TNM classification including downstaged tumor based on adequate imaging of the thorax and abdomen;
4. Intention for right hemicolectomy (including extended right hemicolectomy) with primary anastomosis;
5. Informed consent according to local requirements Exclusion criteria

1) T4b tumor determined by CT scan; 2) Malignancy other than adenocarcinoma at histological examination ; 3)Other malignancies in medical history, except adequately treated basocellular carcinoma of the skin or in situ carcinoma of the cervix uteri; 4) Previous history of colorectal cancer or synchronous multiple colorectal malignancies; 5) Complications requiring emergency surgery (obstruction, perforation, etc); 6) Planned synchronous abdominal organ resections; 7) Pregnant or lactating women; 8) Familial Adenomatosis Polyposis Coli (FAP), active Crohn's disease or active ulcerative colitis; 9) Absolute contraindication to general anesthesia or laparoscopic surgery.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1158 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
Anastomotic leak | 30 days
  Anastomotic leakage is defined as a defect of the intestinal wall at the anastomotic site leading to a communication between intra- and extraluminal compartments.
  Diagnosis of anastomotic leakage: The radiological examination (CT abdomen) will be completed if clinically suspected AL. AL is confirmed clinically, radiologically, endoscopically or intraoperatively. The severity of anastomotic leakage was judged with reference to the Clavien-Dindo classification.

SECONDARY OUTCOMES:
Disease-free survival rate | 3/5 years
  Main secondary outcome
Overall survival | 3/5 years
morbidity | 5 years
Mortality | 5 years
Duration of surgery | Intraoperative
  from incision to suture completion
Duration of anastomosis | Intraoperative
  from the start of dissection of the bowel to the compeletion of the anastomosis
Surgical incision length | Intraoperative
Conversion rate | 1 month
  conversion to open surgery or conversion to extracorporeal anastomosis
Pain score (VAS score) | 1-3 days
  The Visual Analogue Scale (VAS) measures pain intensity. The VAS consists of a 10cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be'). Ask the patient to rate their current level of pain by placing a mark on the line.
Time to first flatus passage after surgery | 1 month
  The day of surgery is day 0. The time interval between the day of the first flatus passage after surgery and the day of surgery.
Time to first stool passage after surgery | up to 1 week
  The day of surgery is day 0. The time interval between the day of the first stool passage after surgery and the day of surgery.
Time to first oral intake | up to 1 week
  The day of surgery is day 0. The time interval between the day of the first oral intake after surgery and the day of surgery.
Length of hospital stay after surgery | 1 month
  days from surgery to discharge
Specimen quality | 1 month
  West pathological assessment criteria. Grading of the plane of mesocolic dissection.
  1. Muscularis propria plane：little bulk to mesocolon with disruptions extending down onto the muscularis propriapropria
  2. Intramesocolic plane: moderate bulk to mesocolon with irregularity but the incisions do not reach down to the muscularis propria
  3. Mesocolic plane: intact mesocolon with a smooth peritoneal-lined surface
Health-related quality of life | 1 year
  EORTC QLQ-CR29 and C30: questionnaires to evaluate the overall quality of life of patients with colorectal cancer, including 30 and 29 items, respectively, to score patients' overall quality of life, function, and symptoms. These are coded with four-point scales, namely "Not at all", "A little", "Quite a bit" and "Very much."
health-related quality of life | 1 year
  EQ 5D-5L (Euroqol): This questionnaire is a simple, generic tool for describing and assessing health-related quality of life. It consists of 5 items (mobility, personal care, activities of daily living, pain and anxiety and depression) that answer questions on a 5-point scale ranging from "no problem" (level 1) to "very severe" (level 5).
Incision herniation | 1 year
  The incision herniation is classified by the criteria of the European Hernia Society. The location (Midline/Lateral) and size (length and width) of the herniation will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Zhongtao Zhang, Prof, Principal Investigator — Department of General Surgery, Beijing Friendship Hospital, Capital Medical University; Hendrik J Bonjer, Prof, Principal Investigator — Amsterdam UMC, location VUmc; Hongwei Yao, Prof, Study Director — Department of General Surgery, Beijing Friendship Hospital, Capital Medical University

IPD SHARING:
Plan to Share IPD: No
We are not sharing confidential individual patient data.